CLINICAL TRIAL: NCT07119307
Title: Evaluation of Entire Papilla Preservation Technique in Combination With Enamel Matrix Derivative & Bone Mineral Derived Xenograft in Isolated Interdental Intrabony Defects
Brief Title: Papilla Preservation Technique in Combination With Tooth Enamel Proteins and Animal Derived Bone Graft in Treating Isolated Bone Defects Between Teeth
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rungta College of Dental Sciences and Research (Other)
Responsible Party: Principal Investigator, Karthik Krishna M, Principal Investigator, Rungta College of Dental Sciences and Research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCDSR/IEC/MDS/2023/D-35
Record Dates: First submitted 2025-08-11; First posted 2025-08-13 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2023-05

CONDITIONS: Periodontal Diseases; Intrabony Periodontal Defect
MeSH Terms: conditions — Periodontal Diseases | interventions — Single Person

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Entire Papilla Preservation Technique (Placebo Comparator): Entire Papilla Preservation Technique alone
  Interventions: Procedure: Entire Papilla Preservation Technique
- Entire Papilla Preservation Technique with Emdogain (Active Comparator): Entire Papilla Preservation Technique with Emdogain
  Interventions: Procedure: Entire Papilla Preservation Surgical Technique (EPPT) alone
- Entire Papilla Preservation Technique with Emdogain and Bovine Derived Xenograft (Active Comparator): Entire Papilla Preservation Technique with Emdogain and Bovine Derived Xenograft
  Interventions: Procedure: Entire Papilla Preservation Surgical Technique (EPPT) alone and combined with enamel matrix derivative (EMD)

INTERVENTIONS:
Procedure: Entire Papilla Preservation Technique — Entire Papilla Preservation Surgical Technique (EPPT) alone and combined with enamel matrix derivative (EMD) plus bone mineral derived xenograph (BMDX)
  Arms: Entire Papilla Preservation Technique
Procedure: Entire Papilla Preservation Surgical Technique (EPPT) alone — Entire Papilla Preservation Surgical Technique (EPPT) alone
  Arms: Entire Papilla Preservation Technique with Emdogain
Procedure: Entire Papilla Preservation Surgical Technique (EPPT) alone and combined with enamel matrix derivative (EMD) — Entire Papilla Preservation Surgical Technique (EPPT) alone and combined with enamel matrix derivative (EMD)
  Arms: Entire Papilla Preservation Technique with Emdogain and Bovine Derived Xenograft

SUMMARY:
The present three-arm study compared the clinical and tomographic efficacy of the Entire Papilla Preservation Surgical Technique (EPPT) alone and combined with enamel matrix derivative (EMD) plus bone mineral derivedxenograph (BMDX), in the treatment of isolated, inter-dental intra-bony defects.

DETAILED DESCRIPTION:
This randomized controlled clinical and tomographic study included 48 sites with isolated interdental intrabony defects, divided into three groups. Group 1 (control) received EPPT alone, Group 2 received EPPT with EMD, and Group 3 received EPPT with EMD and BMDX (Fix-Oss xenograft). Clinical parameters probing pocket depth (PPD), relative attachment level (RAL), gingival recession (GR), and papilla height-were recorded at baseline and 12 months. Cone-beam computed tomography (CBCT) was used to evaluate tomographic changes including defect width, CEJ-BD, CEJ-AC, X-ray INFRA and defect angle.

ELIGIBILITY:
Inclusion Criteria:

* stage II or III periodontitis, according to WWP 2017 classification of periodontal diseases in need of periodontal regenerative treatment for isolated intrabony defects
* single-rooted teeth/multi-rooted teeth without furcation involvement

Exclusion Criteria:

* uncontrolled or poorly controlled diabetes,
* unstable or life-threatening conditions, or requiring antibiotic prophylaxis,
* History of use of medications since last 6 months (immunosuppressants and antibiotics),
* Subjects allergic to medications,
* Pregnant or lactating women, Smokers/users of other tobacco products,
* Subjects showing unacceptable oral hygiene maintenance after initial phase I therapy and
* multiple interconnected vertical defects.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
relative attachment level gain | 6 months
  measuring relative attachment level gain with UNC-15 probe
pocket depth change | 6 months
  measuring probing pocket depth changes

SECONDARY OUTCOMES:
Tomographic defect width | 6 months
  measured defect width in CBCT
the distance between the cemento-enamel junction and the bottom of the defect | 6 months
  the distance between the cemento-enamel junction and the bottom of the defect

CONTACTS AND LOCATIONS:
Locations (1):
- Rungta College of Dental Sciences and Research, Bhilai, Chhattisgarh, India

IPD SHARING:
Plan to Share IPD: Undecided
For confidentiality

REFERENCES:
- [Background] Aslan S, Buduneli N, Cortellini P. Entire Papilla Preservation Technique: A Novel Surgical Approach for Regenerative Treatment of Deep and Wide Intrabony Defects. Int J Periodontics Restorative Dent. 2017 Mar/Apr;37(2):227-233. doi: 10.11607/prd.2584. PMID 28196163